CLINICAL TRIAL: NCT06934681
Title: Impact of a Structured Physical Exercise Program on Body Composition in Morbid Obesity: A Randomized Controlled Trial
Brief Title: Exercise to Fight Obesity
Acronym: ExFO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: University of Valencia (Other); Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Paolo Rossetti, Clinical Researcher, Instituto de Investigacion Sanitaria La Fe
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-1010-1
Record Dates: First submitted 2025-03-30; First posted 2025-04-18 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Morbid Obesity; Bariatric Surgery; Telerehabilitation
Keywords: Bariatric surgery; Physical Exercise; Telerehabilitation; Prehabilitation; Rehabilitation; Body composition; Morbid obesity; Functional capacity
MeSH Terms: conditions — Obesity, Morbid; Motor Activity | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: This is a randomized, pragmatic, superiority clinical trial with two parallel groups (1:1 ratio), conducted with participants diagnosed with obesity who are eligible for bariatric surgery (BS). Eligible participants who consent to participate will be randomly assigned to either a structured physical exercise (PE) program consisting of supervised strength training with a physiotherapist and telerehabilitation-based strength and aerobic sessions combined with physical activity (PA) promotion, or to the standard care protocol currently implemented at the hospital, which includes general guidance on physical activity, exercise, and nutrition. Both groups will receive the same nutritional intervention.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Eligible participants who consent to participate will be randomly assigned to either the standard care group or a physical exercise (PE) program incorporating telerehabilitation. Randomization will be performed using permuted blocks of six participants to ensure balanced allocation and concealment. The randomization sequence will be generated by an independent researcher not involved in participant recruitment or group assignment, and will be concealed in sequentially numbered, opaque, and sealed envelopes.
  After the baseline assessment, study personnel will open the next envelope in the sequence, and the assigned intervention will commence immediately. To preserve methodological rigor, both the evaluators conducting participant assessments and the researchers performing data analyses will remain blinded to group allocation throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided physical exercise with telerehabilitation (Experimental): Participants will engage in structured physical exercises, including both aerobic and strength training, guided and monitored by physiotherapists. These exercises will be performed both in person and remotely with the support of telerehabilitation.
  Interventions: Behavioral: Controlled exercise with telerehabilitation
- Common physical exercise recommendations given in routine clinical practice (Active Comparator): Participants will receive the usual dietary and physical activity recommendations during medical assessments and group sessions.
  Interventions: Behavioral: Usual Care Group

INTERVENTIONS:
Behavioral: Usual Care Group — Participants will receive the standard intervention provided by the healthcare service, which includes recommendations for physical exercise, physical activity, and healthy eating. This intervention is delivered by the Endocrinology and Nutrition Department at Hospital Universitario y Politécnico La Fe and consists of periodic individual follow-ups (at least three in-person visits per year, both pre- and post-bariatric surgery) by specialized medical staff in Endocrinology and licensed Nutrition and Dietetics professionals. Additionally, it includes five preoperative group sessions focusing on various aspects of healthy nutrition, physical exercise, and physical activity.
  Arms: Common physical exercise recommendations given in routine clinical practice
Behavioral: Controlled exercise with telerehabilitation — Participants will receive the same standard care as the control group, including the same number of visits with the physician and nutritionist and participation in group sessions. Additionally, they will follow a structured physical exercise program, tailored to individual capabilities, combining aerobic and strength exercises, which will primarily be carried out at home with the assistance of telerehabilitation. Physical exercise will be structured in different phases: prior to surgery (prehabilitation), after surgery (rehabilitation), with maintenance periods in between.
  Arms: Guided physical exercise with telerehabilitation

SUMMARY:
This clinical trial aims to determinate whether a structured exercise program, supported by telerehabilitation, can help individuals with severe obesity who are going to undergo bariatric surgery.

The main objective of this study is whether a structured exercise program, including both supervised and home-based workouts, leads to greater body fat loss and improved strength compared to usual care. Furthermore, it also aims to evaluate other potentially affected aspects, such as body composition and functionality, quality of life, cardiovascular fitness, and various genetic and metabolic factors.

This study is a randomized clinical trial with two groups:

* The intervention group will follow a structured exercise program both pre- and post- surgery.
* The control group will receive standard care, including nutritional counseling and general health advice.

The study will include 72 adults with severe obesity (36 men and 36 women), all of whom will be randomly assigned to either the intervention or control group.

Participants in the exercise group will follow these steps:

1. Before Surgery (Prehabilitation): A 26-week program with aerobic and strength exercises, done in-person or remotely 2-4 times per week.
2. Pre-Surgery Maintenance: A flexible period before surgery where participants continue exercising on their own.
3. After Surgery (Rehabilitation): A 20-week program focused on recovery and strength.
4. Post-Surgery Maintenance: A long-term, self-guided phase to maintain progress.

Participants in the exercise group will also receive the same care as the control group, including nutrition counseling and medical checkups.

To evaluate participant progress, a series of measurements will be carried out, including:

* BMI and body composition
* Physical function assessed through isometric strength tests and other measures such as the Sit-to-Stand test and the 6-Minute Walk Test
* Quality of life and lifestyle assessed using validated questionnaires
* Daily physical activity measured with pedometers
* Metabolic and genetic analysis from blood samples

If proven effective, this program could help establish structured exercise with telerehabilitation as a standard component of obesity care. The results may support the integration of exercise programs into clinical practice, leading to improved long-term outcomes for individuals with severe obesity undergoing bariatric surgery. Additionally, insights into genetic and metabolic factors may contribute to the development of personalized treatment strategies.

DETAILED DESCRIPTION:
INTRODUCTION Severe obesity represents a growing public health challenge in Spain, with a marked increase in prevalence and significant implications for morbidity, mortality, and healthcare expenditure. In 2022, nearly 400,000 individuals were affected by class III obesity, reflecting an increase of more than 200% since the 1990s. This condition is strongly associated with serious comorbidities, including cardiovascular disease, type 2 diabetes, and certain cancers, and is linked to a substantial reduction in life expectancy. From an economic perspective, overweight and obesity are estimated to account for approximately 10% of national healthcare costs, with severe obesity contributing significantly through both direct medical expenses and indirect costs related to productivity loss.

Conventional treatment strategies, such as dietary interventions and physical activity (PA), offer limited long-term effectiveness in individuals with severe obesity. Although physical exercise (PE)-a structured form of PA-has shown benefits beyond weight reduction, including improvements in body composition and cardiorespiratory fitness, the majority of participants find it difficult to sustain behavioral changes over time. Furthermore, the degree of weight loss required in this population frequently exceeds what lifestyle interventions alone can achieve.

Bariatric surgery has emerged as an effective alternative, providing substantial short-term weight reduction and improvement in obesity-related comorbidities. However, it is not without limitations, including the loss of lean body mass and the risk of long-term weight regain, particularly in the absence of adequate PA following surgery. Recent studies have shown that postoperative PE programs may improve these outcomes, although the evidence on the benefits of preoperative exercise (prehabilitation) remains limited.

In this context, telerehabilitation appears to be a promising strategy for enhancing accessibility, adherence, and continuity of care. Remote supervision of structured exercise programs, supported by wearable technologies such as activity trackers, may help overcome common barriers and increase participant engagement. Additionally, the substantial variability in individual responses to obesity treatment highlights the need for personalized interventions. Genetic, metabolic, and epigenetic factors likely contribute to treatment resistance in certain individuals, and the identification of predictive biomarkers may help guide more effective and individualized obesity management strategies.

OBJECTIVES:

Primary Objective To evaluate whether a structured PE and PA promotion program, incorporating both supervised in-person and home-based sessions through telerehabilitation tools, is more effective than standard care guidelines in reducing fat percentage and increasing lower-limb strength in candidates for bariatric surgery.

Secondary Objectives

To determine whether the structured PE and PA program is more effective than standard care in achieving:

1. Improved physical functionality.
2. Greater cardiovascular capacity.
3. Enhanced quality of life.
4. Superior outcomes in other body composition variables.

Additional secondary objectives include:

1. Evaluating adherence to the recommended session frequency and prescribed training volume.
2. Analyzing the relative contribution, adjusted for sex, of fat percentage reduction and lower-limb strength improvement to functionality and quality of life.
3. Assessing the effects of the PE and PA program on plasma levels of adipokines, exerquines, and cytokines.
4. Investigating epigenetic modifications induced by the PE program.
5. Identifying differences in metabolic, genetic, and epigenetic profiles according to physical fitness level and total volume of PE and PA performed (stratified by activity level, independent of group allocation).
6. Exploring associations between body composition and functional variables with metabolic, genetic, and epigenetic factors.

METHODOLOGY The methodology of the study is included in the initial summary and detailed in the subsequent sections (study design, arms and interventions, outcomes measures and elegibility) .

SAMPLE SIZE The sample size for this clinical trial was determined based on the two coprimary outcomes: fat percentage and lower-limb strength. For fat percentage, the calculation aimed to detect a 2% reduction in the experimental group compared to the control group, with 80% statistical power and a 5% significance level, resulting in an estimated minimum of 13 participants per group. Similarly, for lower-limb strength, assessed via the 5-repetition Sit-to-Stand (5STS) test, a 30% improvement was considered clinically relevant, requiring only 6 participants per group under the same statistical assumptions.

Given that the variable with the higher sample size requirement was fat percentage, it was used to guide the final sample size. To allow for subgroup analyses by sex, the study was designed to include 30 participants per group-15 women and 15 men. To accommodate an anticipated dropout rate of 20%, the final sample size was increased to 36 participants in each group, with equal sex distribution (18 women and 18 men per group).

STATISTICAL METHODS Data management and statistical analyses will be performed using SPSS software. A dedicated study database will be created, and data accuracy will be verified through random cross-checks with original records. Prior to analysis, data cleaning will be conducted to ensure consistency and completeness, followed by the creation of derived variables where necessary.

The analysis will begin with a flowchart of participant progression throughout the study, alongside a comparison of baseline characteristics between groups to assess equivalence at enrollment. Descriptive statistics will be used: categorical variables will be reported as frequencies and percentages, while continuous variables will be expressed as means and standard deviations or medians and interquartile ranges, depending on data distribution.

To evaluate the primary outcomes, a mixed-model ANOVA will be conducted, with time (baseline, end of prehabilitation, and pre-surgery) as the within-subject factor and group allocation (intervention vs. control) as the between-subject factor. The assumptions of normality and homogeneity will be tested using the Shapiro-Wilk and Levene's tests, respectively. When assumptions are violated, appropriate statistical corrections will be applied.

Effect sizes will be reported using partial eta squared (η²), and post hoc analyses will include Bonferroni correction when significant group-time interactions are detected. The magnitude of observed effects will be interpreted using Cohen's d.

The same statistical approach will be applied to secondary outcomes, such as physical function, cardiovascular fitness, quality of life, and body composition. Intervention adherence will be quantified by the proportion of completed sessions and those performed at the prescribed intensity, followed by between-group comparisons using non-parametric tests as appropriate.

To assess the influence of fat mass reduction and improved lower-limb strength on clinically relevant outcomes (e.g., Six-Minute Walk Test [6MWT], Impact of Weight on Quality of Life [IWQOL]), participants will be dichotomized based on whether they achieved a minimally clinically important difference. Multivariate logistic regression models will be constructed, using these two variables and sex as predictors. Model refinement will be carried out via backward elimination, and results will be presented as odds ratios with 95% confidence intervals.

Finally, linear regression models will be used to explore associations between body composition and functional outcomes with genetic, metabolic, and epigenetic markers.

SUBSTUDY 2: POSTOPERATIVE REHABILITATION FOLLOWING BARIATRIC SURGERY In addition to the main study, a subgroup of participants will be enrolled exclusively in the postoperative phase, forming part of Substudy 2. This substudy targets individuals already on the bariatric surgery waiting list and focuses solely on postoperative rehabilitation and maintenance.

The study design and intervention protocols are identical to those of the main study, but the follow-up period is limited to 12 months. Measurements will be conducted at three time points: prior to surgery, 6 months post-surgery, and 12 months post-surgery.

The key differences between the two substudies are as follows:

* Primary Outcome Measures: Given the exclusive postoperative focus of Substudy 2, the primary endpoints differ from those in the main study:

  * Lean Mass Reduction: Assessed via bioelectrical impedance analysis (BIA), this outcome is prioritized over fat percentage reduction, as substantial fat mass loss is expected in all participants following surgery.
  * Lower-Limb Strength: Evaluated using the Five-Repetition Sit-to-Stand (5STS) test, which serves as a functional indicator of muscular performance and recovery.
* Sample Size: The sample size was calculated to detect a directional hypothesis of a 25% smaller decrease in lean mass in the experimental group compared to the control group (effect size f = 0.8), with 80% power and a 5% significance level. This calculation yielded a minimum requirement of 15 participants per group.

To allow for sex-based subgroup analyses, each group (intervention and control) must include 30 participants-15 women and 15 men. Considering an expected dropout rate of approximately 15% in this substudy, the final sample size will be increased to 34 participants per group, resulting in a total of 68 participants overall.

Aside from the differences outlined above, all remaining aspects of Substudy 2-including methodology, intervention content, and assessment procedures-will follow the same protocols described in the main study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* BMI ≥35 with comorbidities, or ≥40, regardless of comorbidity presence

Exclusion Criteria:

* Participation in a structured physical exercise program within the past 6 months
* Presence of musculoskeletal or systemic diseases that prevent participation in a physical exercise program
* Uncontrolled hypertension
* Uncontrolled diabetes, particularly in the presence of severe complications (neuropathy and/or diabetic foot, proliferative retinopathy)
* Uncontrolled or unstable cardiovascular disease (acute myocardial infarction within the past year, angina, heart failure, peripheral artery disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Fat mass percentage | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  The percentage of fat mass relative to the patient's total body mass, measured using bioelectrical impedance analysis (BIA).
Lower limb strength | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  Measured by the 5 repetitions Sit-To-Stand test (5STS)

SECONDARY OUTCOMES:
Weight | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  Measured with BIA machine. Units: kilograms
Height | Baseline
  Measured using a stadiometer permanently fixed to a wall to minimize variability between patients.
  Units: meters
Waist circumference | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  Measured with a non-elastic tape measure. Units: centimeters
Skeletal muscle mass | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  Measured using bioelectrical impedance analysis (BIA).
Lean body mass | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  Measured using bioelectrical impedance analysis (BIA).
Visceral fat area | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  Measured using bioelectrical impedance analysis (BIA).
Blood preasure | Baseline, 6 months, perioperative, 6 moths after and 1 year after
Isometric muscle strength | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  Measured with hand grip, knee extension and elbow flexion. Units: kilograms
6 minutes walking test (6MWT) | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  The 6WMT measures the distance the patient travels in 6 minutes walking as fast as they can.
  The total distance walked is recorded in meters. The greater the distance, the better the results.
Short Performance Physical Battery (SPPB) | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  The SPPB consists of three components:
  * Balance tests:: The participant is asked to maintain balance in three positions: side-by-side stance, semi-tandem stance, and full tandem stance, each for up to 10 seconds.
  * Speed test: The time taken to walk 4 meters
  * Chair stand test: The participant is instructed to stand up and sit down from a chair five times as quickly as possible without using their arms. The time taken is recorded.
  Each component is scored from 0 to 4 points, with a maximum total score of 12. Higher scores indicate better physical performance. The SPPB is widely used in clinical and research settings for assessing frailty, risk of disability, and physical function.
VO2max/VO2 peak | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  Estimated through 6MWT
Steps per day | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  We will provide patients with pedometers to monitor their daily mobility.
International Physical Activity Questionnaire (IPAQ): | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  The IPAQ collects information on physical activity performed in the last 7 days across three specific types: walking, moderate-intensity activities and vigorous-intensity activities.
  Participants are asked to report the frequency (days per week) and duration (minutes per day) of each activity type. The questionnaire also includes a question on time spent sitting, to estimate sedentary behavior.
  Physical activity data are converted into Metabolic Equivalent of Task (MET)-minutes/week, allowing categorization of individuals into three levels of physical activity: low, moderate, or high.
International Sedentary Assessment Tool (ISAT) | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  Participants report the average amount of time spent in sedentary behaviors on a typical weekday and weekend day. The questions activities analyze the time spent sitting while doing some activities such as working, transportation, watching television or using screens.
Short Form-36 Health Survey (SF-36) | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  It evaluates eight dimensions of health across physical and mental domains: Physical Function, Physical Role; Bodily Pain; General Health; Vitality; Social Function; Emotional Role and Mental Health.
  Each dimension is scored from 0 to 100, with higher scores indicating better health status.
Impact of Weight on Quality of Life (IWQOL) | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  It evaluates the physical, emotional, and social impact of overweight and obesity on daily functioning and well-being. It's grouped into five domains: physical function, self-esteem, sexual life, public distress and work.
  Participants rate how true each statement is for them, using a 5-point scale. Minimum value: 31, Maximum value: 155 Higher scores indicate better weight-related quality of life.
Bariatric Analysis and Reporting Outcome System (BAROS) | 6 months post-surgery and one year post-surgery.
  The BAROS assesses different aspects of patients undergoing bariatric surgery, including the percentage of excess weight lost, comorbidities and quality of life.
  Each domain is scored and higher scores indicate better outcomes. Minimum value: 0, Maximum value: 48
Number of participants with abnormal laboratory tests results | Baseline, 6 months, perioperative, 6 moths after and 1 year after
  Several analytical parameters will be assessed in the participants, including complete blood count, biochemical analysis with electrolytes, renal and hepatic function, glycemic levels and HbA1c, albumin levels, vitamin profile, and markers of iron metabolism. Furthermore, the quantification of various exerkines, adipokines, and cytokines will also be conducted.
Number of participants with genetic alterations | Baseline (Stored in a biobank for analysis if funding is obtained)
  A genetic panel targeting obesity-related genes will be performed if funding is secured. Initially, the samples will be stored in a biobank. The following exons will be analyzed:
  ABCC8, ACBD6, ADCY3, ADRB2, AFF4, AKR1C2, ALMS1, ARL6, BBIP1, BBS1, BBS10, BBS12, BBS2, BBS4, BBS5, BBS7, BBS9, BDNF, CEL, CEP164, CEP19, CEP290, CPE, CREBBP, CUL4B, CYP27A1, DNMT3A, DYRK1B, EHMT1, EIF2AK3, ENPP1, EP300, FOXP3, FTO, GCK, GHRL, GLIS3, GNAS, GNB1, HNF1A, HNF1B, HNF4A, IFNGR1, IFT172, IFT27, IFT74, INPP5E, INS, KCNJ11, KDM6A, KIDINS220, KIF7, KMT2D, KSR2, LEP, LEPR, LZTFL1, MAGEL2, MC4R, MEGF8, MKKS, MKRN3, MKS1, MRAP2, MYT1L, NDN, NEUROD1, NEUROG3, NLGN2, NR0B2, NTRK2, P4HTM, PCSK1, PDE4D, PDX1, PGM2L1, PHF6, PHIP, POMC, PPARG, PRKAR1A, PRKN, PRMT7, PTF1A, RAB23, RAD21, RAI1, RFX6, RPS6KA3, SCAPER, SCLT1, SDCCAG8, SETD1B, SETD2, SH2B1, SIM1, SNRPN, STX16, TFAP2B, TMEM67, TRAPPC9, TRIM32, TTC8, TUB, VPS13B, WDPCP, WFS1.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Rossetti, Medicine, Principal Investigator — IIS La Fe; Rodrigo Martín, Study Director — Grupo de investigación Clinimetría y desarrollo tecnológico en ejercicio terapéutico (CLIDET); Pilar Masdeu, Medicine, Study Chair — IIS La Fe; Noemí Moreno, Study Chair — CLIDET; Ana Belén Crujeiras, Study Chair — Unidad de Epigenómica en el Instituto de Investigación Sanitaria de Santiago (IDIS); Maria Dolores Herranz Lopez, Study Chair — Universidad Miguel Hernández; Adrián Escriche, Study Chair — CLIDET; Cristina Flor, Study Chair — CLIDET; Albert Lecube, Study Chair — Sociedad Española para el Estudio de la Obesidad (SEEDO); Enrique Roche Collado, Study Chair — Universidad Miguel Hernández
Locations (2):
- Spain (2):
  - Facultad de Fisioterapia, universidad de Valencia, Valencia, Valencia
  - Hospital La Fe, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Brien PE, Sawyer SM, Laurie C, Brown WA, Skinner S, Veit F, Paul E, Burton PR, McGrice M, Anderson M, Dixon JB. Laparoscopic adjustable gastric banding in severely obese adolescents: a randomized trial. JAMA. 2010 Feb 10;303(6):519-26. doi: 10.1001/jama.2010.81. PMID 20145228
- [Background] Must A, Spadano J, Coakley EH, Field AE, Colditz G, Dietz WH. The disease burden associated with overweight and obesity. JAMA. 1999 Oct 27;282(16):1523-9. doi: 10.1001/jama.282.16.1523. PMID 10546691
- [Background] Marc-Hernandez A, Ruiz-Tovar J, Aracil A, Guillen S, Moya-Ramon M. Impact of Exercise on Body Composition and Cardiometabolic Risk Factors in Patients Awaiting Bariatric Surgery. Obes Surg. 2019 Dec;29(12):3891-3900. doi: 10.1007/s11695-019-04088-9. PMID 31313237
- [Background] Loveman E, Frampton GK, Shepherd J, Picot J, Cooper K, Bryant J, Welch K, Clegg A. The clinical effectiveness and cost-effectiveness of long-term weight management schemes for adults: a systematic review. Health Technol Assess. 2011 Jan;15(2):1-182. doi: 10.3310/hta15020. PMID 21247515
- [Background] Li J, Lin Y, Deng H, Su X, Feng W, Shao Q, Zou K. Association of visceral adiposity index with sarcopenia based on NHANES data. Sci Rep. 2024 Sep 10;14(1):21169. doi: 10.1038/s41598-024-72218-0. PMID 39256533
- [Background] Levitt DG, Beckman LM, Mager JR, Valentine B, Sibley SD, Beckman TR, Kellogg TA, Ikramuddin S, Earthman CP. Comparison of DXA and water measurements of body fat following gastric bypass surgery and a physiological model of body water, fat, and muscle composition. J Appl Physiol (1985). 2010 Sep;109(3):786-95. doi: 10.1152/japplphysiol.00278.2010. Epub 2010 Jun 17. PMID 20558754
- [Background] Karmali S, Brar B, Shi X, Sharma AM, de Gara C, Birch DW. Weight recidivism post-bariatric surgery: a systematic review. Obes Surg. 2013 Nov;23(11):1922-33. doi: 10.1007/s11695-013-1070-4. PMID 23996349
- [Background] Jensen SBK, Blond MB, Sandsdal RM, Olsen LM, Juhl CR, Lundgren JR, Janus C, Stallknecht BM, Holst JJ, Madsbad S, Torekov SS. Healthy weight loss maintenance with exercise, GLP-1 receptor agonist, or both combined followed by one year without treatment: a post-treatment analysis of a randomised placebo-controlled trial. EClinicalMedicine. 2024 Feb 19;69:102475. doi: 10.1016/j.eclinm.2024.102475. eCollection 2024 Mar. PMID 38544798
- [Background] Jabbour G, Ibrahim R, Bragazzi N. Preoperative Physical Activity Level and Exercise Prescription in Adults With Obesity: The Effect on Post-Bariatric Surgery Outcomes. Front Physiol. 2022 Jul 6;13:869998. doi: 10.3389/fphys.2022.869998. eCollection 2022. PMID 35874538
- [Background] Huck CJ. Effects of supervised resistance training on fitness and functional strength in patients succeeding bariatric surgery. J Strength Cond Res. 2015 Mar;29(3):589-95. doi: 10.1519/JSC.0000000000000667. PMID 25226310
- [Background] Hassannejad A, Khalaj A, Mansournia MA, Rajabian Tabesh M, Alizadeh Z. The Effect of Aerobic or Aerobic-Strength Exercise on Body Composition and Functional Capacity in Patients with BMI >/=35 after Bariatric Surgery: a Randomized Control Trial. Obes Surg. 2017 Nov;27(11):2792-2801. doi: 10.1007/s11695-017-2717-3. PMID 28527156
- [Background] Hansen BH, Holme I, Anderssen SA, Kolle E. Patterns of objectively measured physical activity in normal weight, overweight, and obese individuals (20-85 years): a cross-sectional study. PLoS One. 2013;8(1):e53044. doi: 10.1371/journal.pone.0053044. Epub 2013 Jan 7. PMID 23308135
- [Background] Global BMI Mortality Collaboration, Di Angelantonio E, Bhupathiraju ShN, Wormser D, Gao P, Kaptoge S, Berrington de Gonzalez A, Cairns BJ, Huxley R, Jackson ChL, Joshy G, Lewington S, Manson JE, Murphy N, Patel AV, Samet JM, Woodward M, Zheng W, Zhou M, Bansal N, Barricarte A, Carter B, Cerhan JR, Smith GD, Fang X, Franco OH, Green J, Halsey J, Hildebrand JS, Jung KJ, Korda RJ, McLerran DF, Moore SC, O'Keeffe LM, Paige E, Ramond A, Reeves GK, Rolland B, Sacerdote C, Sattar N, Sofianopoulou E, Stevens J, Thun M, Ueshima H, Yang L, Yun YD, Willeit P, Banks E, Beral V, Chen Zh, Gapstur SM, Gunter MJ, Hartge P, Jee SH, Lam TH, Peto R, Potter JD, Willett WC, Thompson SG, Danesh J, Hu FB. Body-mass index and all-cause mortality: individual-participant-data meta-analysis of 239 prospective studies in four continents. Lancet. 2016 Aug 20;388(10046):776-86. doi: 10.1016/S0140-6736(16)30175-1. Epub 2016 Jul 13. PMID 27423262
- [Background] Dixon JB, O'Brien PE, Playfair J, Chapman L, Schachter LM, Skinner S, Proietto J, Bailey M, Anderson M. Adjustable gastric banding and conventional therapy for type 2 diabetes: a randomized controlled trial. JAMA. 2008 Jan 23;299(3):316-23. doi: 10.1001/jama.299.3.316. PMID 18212316
- [Background] Dent R, McPherson R, Harper ME. Factors affecting weight loss variability in obesity. Metabolism. 2020 Dec;113:154388. doi: 10.1016/j.metabol.2020.154388. Epub 2020 Oct 7. PMID 33035570
- [Background] Coleman KJ, Caparosa SL, Nichols JF, Fujioka K, Koebnick C, McCloskey KN, Xiang AH, Ngor EW, Levy SS. Understanding the Capacity for Exercise in Post-Bariatric Patients. Obes Surg. 2017 Jan;27(1):51-58. doi: 10.1007/s11695-016-2240-y. PMID 27229736
- [Background] Coldebella B, Armfield NR, Bambling M, Hansen J, Edirippulige S. The use of telemedicine for delivering healthcare to bariatric surgery patients: A literature review. J Telemed Telecare. 2018 Dec;24(10):651-660. doi: 10.1177/1357633X18795356. PMID 30343656
- [Background] Clinical Guidelines on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults--The Evidence Report. National Institutes of Health. Obes Res. 1998 Sep;6 Suppl 2:51S-209S. No abstract available. PMID 9813653
- [Background] Chaston TB, Dixon JB, O'Brien PE. Changes in fat-free mass during significant weight loss: a systematic review. Int J Obes (Lond). 2007 May;31(5):743-50. doi: 10.1038/sj.ijo.0803483. Epub 2006 Oct 31. PMID 17075583
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Bruno DS, Berger NA. Impact of bariatric surgery on cancer risk reduction. Ann Transl Med. 2020 Mar;8(Suppl 1):S13. doi: 10.21037/atm.2019.09.26. PMID 32309417
- [Background] Boppre G, Borges LPSL, Diniz-Sousa F, Veras L, Devezas V, Preto J, Santos-Sousa H, da Costa THM, Oliveira J, Fonseca H. Effects of a supervised exercise training on body composition after bariatric surgery: a randomized controlled trial. Obesity (Silver Spring). 2023 Nov;31(11):2750-2761. doi: 10.1002/oby.23894. PMID 37853990
- [Background] Bojarczuk A, Egorova ES, Dzitkowska-Zabielska M, Ahmetov II. Genetics of Exercise and Diet-Induced Fat Loss Efficiency: A Systematic Review. J Sports Sci Med. 2024 Mar 1;23(1):236-257. doi: 10.52082/jssm.2024.236. eCollection 2024 Mar. PMID 38455434
- [Background] Berthoud HR, Munzberg H, Morrison CD. Blaming the Brain for Obesity: Integration of Hedonic and Homeostatic Mechanisms. Gastroenterology. 2017 May;152(7):1728-1738. doi: 10.1053/j.gastro.2016.12.050. Epub 2017 Feb 10. PMID 28192106
- [Background] Bellicha A, van Baak MA, Battista F, Beaulieu K, Blundell JE, Busetto L, Carraca EV, Dicker D, Encantado J, Ermolao A, Farpour-Lambert N, Pramono A, Woodward E, Oppert JM. Effect of exercise training before and after bariatric surgery: A systematic review and meta-analysis. Obes Rev. 2021 Jul;22 Suppl 4(Suppl 4):e13296. doi: 10.1111/obr.13296. Epub 2021 Jun 3. PMID 34080281
- [Background] Basterra-Gortari FJ, Beunza JJ, Bes-Rastrollo M, Toledo E, Garcia-Lopez M, Martinez-Gonzalez MA. [Increasing trend in the prevalence of morbid obesity in Spain: from 1.8 to 6.1 per thousand in 14 years]. Rev Esp Cardiol. 2011 May;64(5):424-6. doi: 10.1016/j.recesp.2010.06.010. Epub 2011 Mar 15. Spanish. PMID 21411209
- [Background] Barbat-Artigas S, Pinheiro Carvalho L, Rolland Y, Vellas B, Aubertin-Leheudre M. Muscle Strength and Body Weight Mediate the Relationship Between Physical Activity and Usual Gait Speed. J Am Med Dir Assoc. 2016 Nov 1;17(11):1031-1036. doi: 10.1016/j.jamda.2016.06.026. Epub 2016 Aug 21. PMID 27553472
- [Background] Anderson JW, Konz EC, Frederich RC, Wood CL. Long-term weight-loss maintenance: a meta-analysis of US studies. Am J Clin Nutr. 2001 Nov;74(5):579-84. doi: 10.1093/ajcn/74.5.579. PMID 11684524